CLINICAL TRIAL: NCT02092389
Title: Fecal Calprotectin Levels, Quality of Life and Workability in Patients Suffering From Ulcerative Colitis Under Adalimumab Therapy - AdaProQuo
Brief Title: Fecal Calprotectin Levels, Quality of Life, and Workability in Patients Suffering From Ulcerative Colitis Under Adalimumab Therapy - AdaProQuo
Acronym: AdaProQuo
Status: Terminated | Type: Observational
Why Stopped: Recruitment below expectation
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-323
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Moderate to Severe Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Syndrome; Adalimumab; Tumor necrosis factor (TNF) alpha Antibody; Calprotectin
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate to Severe Ulcerative Colitis: Patients with moderate to severe ulcerative colitis (UC) who have not responded despite a full and adequate course of therapy with a corticosteroid and an immunosuppressant (azathioprine [AZA]/ 6-mercaptopurine [6-MP]); or who are intolerant to or have medical contraindications for such therapies and are hence prescribed adalimumab for the treatment of moderate to severely active UC.

SUMMARY:
The objectives of this study are to explore the fecal calprotectin (fC) levels of UC patients under adalimumab therapy and the correlation with their general wellbeing (Quality of Life [QoL]), workability, and disease activity.

DETAILED DESCRIPTION:
This is a non-interventional, observational study in which Humira (adalimumab) is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. The assignment of the patient to a adalimumab containing regimen has to be decided in advance and has to be current practice. The prescription of adalimumab is clearly separated from the decision to include the participant in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe ulcerative colitis (UC) who have not responded despite a full and adequate course of therapy with a corticosteroid and an immunosuppressant (AZA/6-MP); or who are intolerant to or have medical contraindications for such therapies and are hence prescribed adalimumab for the treatment of moderate to severely active UC
* Patients who are able to complete patients questionnaires (e.g., WPAI:UC and sIBDQ questionnaire)
* Patients must fulfill national and international guidelines for the use of biologic therapies in UC (Chest X-ray and Interferon-Gamma-Release Assay (IGRA) or tuberculin purified protein derivative (PPD)-skin test negative for tuberculosis).
* Patients who have been prescribed adalimumab in line with the European SmPC (Summary of Product Characteristics)

Exclusion Criteria:

* Previous therapy with TNF-alpha (Tumor necrosis factor alpha) blocker
* No signed written authorization to use data
* Contraindication to adalimumab therapy according to the SmPC
* Patients with a history of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC or planned bowel surgery.
* Patients received intravenous (IV) corticosteroids within 14 days of Screening or during the Screening period.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dorr, MD, Study Director — AbbVie Austria

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate to Severe Ulcerative Colitis
Started | 10
Completed | 4
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants with demographic and baseline data available.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (16.88)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Fecal calprotectin (fC) levels at baseline [Mean (Standard Deviation); unit: μg/g] — fC is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing. fC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. A total of 8 participants had fC baseline data available.
  μg/g | 440 (393.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Fecal Calprotectin (fC) Level ≤ 150 µg/g After 12 Months of Treatment With Adalimumab
Description: Fecal calprotectin (fC) is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing. fC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. The study was terminated due to low enrollment. Although no meaningful analysis can be presented, data for subjects with available data for fC levels at Month 12 at the end of study (termination) are provided.
Time Frame: Month 12
Population: Enrolled participants with Month 12 data at the time of study termination
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 2
percentage of participants | 100

2. Secondary Outcome: Change From Baseline to Month 12 in Patient's Workability Measured Using the Work Productivity and Activity Impairment:Ulcerative Colitis (WPAI:UC) Questionnaire
Description: The WPAI:UC is a questionnaire used to evaluate lost productivity (work time missed and work and activity impairment) during the past 7 days due to UC. The scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Change in WPAI-UC is calculated by deducting the final score from the baseline score. Increased (positive) scores correspond to a reduction in the percentage of lost work productivity.
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline to Month 12 in Patient's Quality of Life (QoL) Measured Using the Short Inflammatory Bowl Disease Questionnaire (sIBDQ)
Description: The sIBDQ is a disease-specific health-related quality of life (QoL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) patients by measuring physical, social and emotional status. The sIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). The scores are summed up and divided by 10 for a mean score ranging from 1 (poor QoL) to 7 (good QoL). Increased scores correspond to an improvement in QoL.
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline to Month 12 in Disease Activity Determined by Partial Mayo Score
Description: A partial mayo score (mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]).
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation Between fC and Disease Activity Determined by Partial Mayo Score
Description: Fecal calprotectin (fC) is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing. fC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. A partial mayo score (mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA).
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation Between fC and Patient's QoL Determined by the sIBDQ
Description: fC is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing. fC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. The sIBDQ is a disease-specific health-related QoL questionnaire, able to detect and define meaningful clinical changes in IBD patients by measuring physical, social and emotional status. The sIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). The scores are summed up and divided by 10 for a mean score ranging from 1 (poor QoL) to 7 (good QoL).
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation Between fC and Workability Determined by WPAI:UC Questionnaire
Description: Fecal calprotectin (fC) is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing. fC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. The WPAI:UC is a questionnaire used to evaluate lost productivity (work time missed and work and activity impairment) during the past 7 days due to UC. The scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline (Day 0) to Month 12
Population: The study was terminated due to low enrollment and data were not collected.
Arm/Group | Moderate to Severe Ulcerative Colitis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time informed consent was obtained until 70 days after the last dose of study drug (up to 14.5 months).
Arm/Group | Moderate to Severe Ulcerative Colitis
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate to Severe Ulcerative Colitis (N=10)
No therapeutic response (General disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated due to low enrollment; therefore, safety and efficacy data should be interpreted with caution because of the small number of participants and incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.